CLINICAL TRIAL: NCT02058589
Title: Observer-blind Study to Evaluate Immunogenicity and Safety of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine GSK1437173A in Adults 18 Years of Age or Older With Renal Transplant
Brief Title: Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine in Adults 18 Years of Age or Older With Renal Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116886; 2012-005059-18 (EudraCT Number)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-06

CONDITIONS: Herpes Zoster
Keywords: Immunocompromised; Safety; ≥ 18 years of age; Renal transplant; Adults; Immunosuppressed; Immunogenicity; Herpes zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK1437173A Group (Experimental): Subjects, aged 18 years or older, received 2 doses of the GSK 1437173A vaccine, adjuvanted with AS01B at Day 0, and Month 1, administered intramuscularly, in the deltoid muscle of an arm.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A
- Placebo Group (Placebo Comparator): Subjects, aged 18 years or older, received 2 doses of Placebo (lyophilised sucrose reconstituted with saline [NaCl] solution) at Day 0, and Month 1, administered intramuscularly, in the deltoid muscle of an arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Herpes Zoster vaccine GSK1437173A — 2 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Arms: GSK1437173A Group
Drug: Placebo — 2 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK Biologicals' HZ/su vaccine administered on a 0- and 1- to 2-months schedule in adults 18 years of age or older who are receiving chronic immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female, aged 18 years or older and having reached the age of legal consent, on the date the informed consent is signed.
* Written informed consent obtained from the subject.
* Subject who has received an ABO compatible allogeneic renal transplant.
* Subject receiving maintenance immunosuppressive therapy for the prevention of allograft rejection for a minimum of one month (30 days) prior to the first vaccination.
* Subject without an episode of allograft rejection over the previous three months (90 days) prior to the first vaccination.
* Subject with stable renal function, stability defined as:

  * less than 20% variability between last two creatinine measurements or calculated GFR
  * or in the opinion of the investigator after investigator review of more than the last two creatinine measurements or calculated GFRs.
* Subject not less than 4 months (120 days) and not more than 18 months (547 days) after allograft transplantation at the time of the first vaccination.
* Subjects with multiple dialysis options (peritoneal and/or more than one anatomical access site for haemodialysis) in the event acute or chronic dialysis is needed.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of the first vaccination, and
  * has agreed to continue adequate contraception during the primary treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Any primary kidney disease with a high incidence of recurrent primary kidney disease.
* Evidence of recurrent primary kidney disease within the current allograft.
* Previous allograft loss secondary to recurrent primary kidney disease.

  * Multiple kidney transplants are allowed if the reason for a previous allograft's loss is not recurrent primary kidney disease.
* More than one organ transplanted (i.e. kidney-liver, double kidney or kidney-other organ(s) transplanted).
* History of events that, in the opinion of the investigator, may put subject at increased risk for chronic allograft dysfunction (e.g. delayed graft function, peri-operative complications).
* Histologic reports of chronic allograft injury (e.g. transplant glomerulopathy, arteriopathy, C4d deposition).
* Evidence of significant proteinuria in the opinion of the investigator.
* Panel reactive antibody score (PRA or cPRA) that is unknown at the time of transplant.
* Any autoimmune or potential immune-mediated disease including primary kidney disease.
* Use of anti-CD20 or other B-cell monoclonal antibody agents (e.g., rituximab) as induction, maintenance and/or therapeutic immunosuppressive therapy for the prevention of allograft rejection within 9 months (274 days) of first dose of study vaccine/placebo.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period.
* Concurrent or planned participation in another clinical study, at any time during the study period, which has exposed or will expose the subject to an investigational or a non-registered product
* Administration or planned administration of a live vaccine within 30 days prior to the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine within 8 days prior to or within 14 days after either dose of study vaccine.
* Planned administration during the study of a varicella or HZ vaccine other than the study vaccine.
* Previous vaccination against HZ or varicella within the 12 months preceding the first dose of study vaccine/placebo.
* Occurrence of varicella or HZ per clinical history, within the 12 months preceding the first dose of study vaccine/placebo.
* Failure to fully complete the 7-day pre-vaccination diary card distributed at the Pre-vaccination visit.
* Evidence or high suspicion, in the opinion of the investigator, of noncompliance or nonadherence to use of induction and/or maintenance immunosuppressive therapies.
* Any confirmed or suspected HIV, primary immunodeficiency disease, disseminated or untreated malignancy, or systemic infection.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine or study material and equipment.
* Any condition which, in the judgment of the investigator, would make intramuscular injection unsafe.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Acute disease and/or fever at the time of vaccination.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F by oral route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) before Month 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
- GSK Investigational Site, Hradec Králové, Czechia
- GSK Investigational Site, Helsinki, Finland
- Italy (5):
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Treviso, Veneto
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Seoul, South Korea
- Spain (7):
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

REFERENCES:
- [Derived] Vink P, Ramon Torrell JM, Sanchez Fructuoso A, Kim SJ, Kim SI, Zaltzman J, Ortiz F, Campistol Plana JM, Fernandez Rodriguez AM, Rebollo Rodrigo H, Campins Marti M, Perez R, Gonzalez Roncero FM, Kumar D, Chiang YJ, Doucette K, Pipeleers L, Aguera Morales ML, Rodriguez-Ferrero ML, Secchi A, McNeil SA, Campora L, Di Paolo E, El Idrissi M, Lopez-Fauqued M, Salaun B, Heineman TC, Oostvogels L; Z-041 Study Group. Immunogenicity and Safety of the Adjuvanted Recombinant Zoster Vaccine in Chronically Immunosuppressed Adults Following Renal Transplant: A Phase 3, Randomized Clinical Trial. Clin Infect Dis. 2020 Jan 2;70(2):181-190. doi: 10.1093/cid/ciz177. PMID 30843046

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 265 subjects originally enrolled in the study, only 264 subjects received vaccination and were hence included in the Total Vaccinated Cohort.
Groups:
- Control Group: Subjects, aged 18 years or older, received 2 doses of Placebo (lyophilised sucrose reconstituted with saline [NaCl] solution) at Day 0, and Month 1, administered intramuscularly, in the deltoid muscle of an arm.
Period: Overall Study
Arm/Group | GSK1437173A Group | Control Group
Started | 132 | 132
Completed | 130 | 130
Not Completed | 2 | 2
Not completed — Serious Adverse Event | 1 | 1
Not completed — Non-Serious Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Control Group | Total
Number analyzed (Participants) | 132 | 132 | 264
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 52.3 (12.5) | 52.4 (12.8) | 52.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 94 | 91 | 185
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 3 | 1 | 4
  Asian - Central/South Asian Heritage | 1 | 2 | 3
  Asian - East Asian Heritage | 20 | 22 | 42
  Asian - Japanese Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 10 | 3 | 13
  White - Arabic / North African Heritage | 2 | 2 | 4
  White - Caucasian / European Heritage | 88 | 97 | 185
  Unspecified | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Vaccine Response for Anti-glycoprotein E (gE) Humoral Immunogenicity
Description: Vaccine response was defined as: For initially seronegative subjects, antibody concentration at post-vaccination greater than or equal to (≥) 4 fold the cut-off for Anti-gE (4x97 milli-international units per milliliter [mIU/ml]); For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration. Vaccine response was determined by Enzyme-Linked ImmunoSorbent Assay (ELISA).
Time Frame: At Month 2.
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for humoral immunogenicity, which included all evaluable subjects up to Month 2, who did not meet any of the criteria for elimination from an ATP analysis, and for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 121 | 119
Participants | 97 | 5

2. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = Pain when limb was moved, which prevented everyday activities. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within 7 days (Days 0-6) after each dose and across doses.
Population: The analysis was performed on the subjects with symptom sheets completed from the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1437173A Group: Subjects, aged 18 years or older, received 2 doses of the GSK 1437173A vaccine, adjuvanted with AS01B at Day 0, and Month 1, administered intramuscularly, in the deltoid muscle of the non-dominant arm.
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 131 | 132
Participants
  Any Pain, Dose 1 | 107 | 8
  Grade 3 Pain, Dose 1 | 10 | 0
  Any Redness, Dose 1 | 24 | 1
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 10 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 125 | 128
  Any Pain, Dose 2 | 93 | 6
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Pain, Dose 2 | 9 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 125 | 128
  Any Redness, Dose 2 | 21 | 1
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 125 | 128
  Any Swelling, Dose 2 | 11 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Swelling, Dose 2 | 1 | 0
  Any Pain, Across doses | 114 | 11
  Grade 3 Pain, Across doses | 13 | 0
  Any Redness, Across doses | 33 | 2
  Grade 3 Redness, Across doses | 1 | 0
  Any Swelling, Across doses | 15 | 1
  Grade 3 Swelling, Across doses | 1 | 0

3. Primary Outcome: Days With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling.
Time Frame: Within 7 days (Days 0-6) after each dose and overall/dose
Population: The analysis was performed on the subjects with solicited local symptoms from the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 114 | 11
Days
  Pain, Dose 1: number analyzed (Participants) | 107 | 8
  Pain, Dose 1 | 3.0 [2.0 to 4.0] | 1.5 [1.0 to 2.5]
  Pain, Dose 2: number analyzed (Participants) | 93 | 6
  Pain, Dose 2 | 3.0 [2.0 to 3.0] | 1.0 [1.0 to 2.0]
  Pain, Overall | 3.0 [2.0 to 4.0] | 1.0 [1.0 to 2.0]
  Redness, Dose 1: number analyzed (Participants) | 24 | 1
  Redness, Dose 1 | 4.0 [2.5 to 6.5] | 4.0 [4.0 to 4.0]
  Redness, Dose 2: number analyzed (Participants) | 21 | 1
  Redness, Dose 2 | 3.0 [2.0 to 7.0] | 2.0 [2.0 to 2.0]
  Redness, Overall: number analyzed (Participants) | 33 | 2
  Redness, Overall | 4.0 [2.0 to 7.0] | 3.0 [2.0 to 4.0]
  Swelling, Dose 1: number analyzed (Participants) | 10 | 1
  Swelling, Dose 1 | 4.0 [2.0 to 7.0] | 4.0 [4.0 to 4.0]
  Swelling, Dose 2: number analyzed (Participants) | 11 | 0
  Swelling, Dose 2 | 4.0 [1.0 to 5.0] |
  Swelling, Overall: number analyzed (Participants) | 15 | 1
  Swelling, Overall | 4.0 [2.0 to 6.0] | 4.0 [4.0 to 4.0]

4. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)] . Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Gastrointestinal symptoms (Gastro. sympt.) included nausea, vomiting, diarrhoea and/or abdominal pain.
Time Frame: Within 7 days (Days 0-6) after each dose and across doses
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Subjects, aged 18 years or older, received 2 doses of Placebo (lyophilised sucrose reconstituted with saline [NaCl] solution) at Day 0, and Month 1, administered intramuscularly, in the deltoid muscle of the non-dominant arm.
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 131 | 132
Participants
  Any Fatigue, Dose 1 | 47 | 42
  Grade 3 Fatigue, Dose 1 | 3 | 3
  Related Fatigue, Dose 1 | 8 | 2
  Any Gastro. sympt., Dose 1 | 17 | 16
  Grade 3 Gastro. sympt., Dose 1 | 1 | 0
  Related Gastro. sympt., Dose 1 | 1 | 1
  Any Headache, Dose 1 | 32 | 25
  Grade 3 Headache, Dose 1 | 1 | 4
  Related Headache, Dose 1 | 5 | 3
  Any Myalgia, Dose 1 | 43 | 23
  Grade 3 Myalgia, Dose 1 | 4 | 1
  Related Myalgia, Dose 1 | 11 | 2
  Any Shivering, Dose 1 | 10 | 13
  Grade 3 Shivering, Dose 1 | 0 | 1
  Related Shivering, Dose 1 | 3 | 2
  Any Temperature, Dose 1 | 13 | 6
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 3 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 125 | 128
  Any Fatigue, Dose 2 | 49 | 36
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Fatigue, Dose 2 | 4 | 4
  Related Fatigue, Dose 2: number analyzed (Participants) | 125 | 128
  Related Fatigue, Dose 2 | 8 | 4
  Any Gastro. sympt., Dose 2: number analyzed (Participants) | 125 | 128
  Any Gastro. sympt., Dose 2 | 14 | 14
  Grade 3 Gastro. sympt., Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Gastro. sympt., Dose 2 | 0 | 1
  Related Gastro. sympt., Dose 2: number analyzed (Participants) | 125 | 128
  Related Gastro. sympt., Dose 2 | 1 | 2
  Any Headache, Dose 2: number analyzed (Participants) | 125 | 128
  Any Headache, Dose 2 | 35 | 22
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Headache, Dose 2 | 2 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 125 | 128
  Related Headache, Dose 2 | 9 | 1
  Any Myalgia, Dose 2: number analyzed (Participants) | 125 | 128
  Any Myalgia, Dose 2 | 47 | 19
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Myalgia, Dose 2 | 8 | 3
  Related Myalgia, Dose 2: number analyzed (Participants) | 125 | 128
  Related Myalgia, Dose 2 | 14 | 3
  Any Shivering, Dose 2: number analyzed (Participants) | 125 | 128
  Any Shivering, Dose 2 | 23 | 9
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Shivering, Dose 2 | 4 | 2
  Related Shivering, Dose 2: number analyzed (Participants) | 125 | 128
  Related Shivering, Dose 2 | 9 | 0
  Any Temperature, Dose 2: number analyzed (Participants) | 125 | 128
  Any Temperature, Dose 2 | 21 | 7
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 125 | 128
  Grade 3 Temperature, Dose 2 | 1 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 125 | 128
  Related Temperature, Dose 2 | 6 | 0
  Any Fatigue, Across doses | 62 | 53
  Grade 3 Fatigue, Across doses | 4 | 6
  Related Fatigue, Across doses | 15 | 4
  Any Gastro. sympt., Across doses | 24 | 24
  Grade 3 Gastro. sympt., Across doses | 1 | 1
  Related Gastro. sympt.,Across doses | 2 | 3
  Any Headache, Across doses | 44 | 34
  Grade 3 Headache, Across doses | 2 | 5
  Related Headache, Across doses | 12 | 4
  Any Myalgia, Dose Across doses | 65 | 31
  Grade 3 Myalgia, Dose Across doses | 9 | 3
  Related Myalgia, Dose Across doses | 21 | 4
  Any Shivering, Dose Across doses | 29 | 16
  Grade 3 Shivering, Dose Across doses | 4 | 2
  Related Shivering, Dose Across doses | 11 | 2
  Any Temperature, Dose Across doses | 31 | 13
  Grade 3 Temperature, Dose Across doses | 1 | 0
  Related Temperature, Dose Across doses | 9 | 0

5. Primary Outcome: Days With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)].
Time Frame: Within 7 days (Days 0-6) after each dose and overall/dose
Population: The analysis was performed on the subjects with solicited general symptoms from the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 65 | 53
Days
  Fatigue, Dose 1: number analyzed (Participants) | 47 | 42
  Fatigue, Dose 1 | 3.0 [2.0 to 6.0] | 3.0 [1.0 to 7.0]
  Fatigue, Dose 2: number analyzed (Participants) | 49 | 36
  Fatigue, Dose 2 | 3.0 [2.0 to 5.0] | 4.5 [2.0 to 7.0]
  Fatigue, Overall: number analyzed (Participants) | 62 | 53
  Fatigue, Overall | 3.0 [2.0 to 5.5] | 4.0 [2.0 to 7.0]
  Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 17 | 16
  Gastrointestinal symptoms, Dose 1 | 2.0 [1.0 to 2.0] | 3.5 [1.0 to 4.5]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 14 | 14
  Gastrointestinal symptoms, Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Gastrointestinal symptoms, Overall: number analyzed (Participants) | 24 | 24
  Gastrointestinal symptoms, Overall | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0]
  Headache, Dose 1: number analyzed (Participants) | 32 | 25
  Headache, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, Dose 2: number analyzed (Participants) | 35 | 22
  Headache, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Headache, Overall: number analyzed (Participants) | 44 | 34
  Headache, Overall | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Myalgia, Dose 1: number analyzed (Participants) | 43 | 23
  Myalgia, Dose 1 | 3.0 [2.0 to 4.0] | 3.0 [1.0 to 7.0]
  Myalgia, Dose 2: number analyzed (Participants) | 47 | 19
  Myalgia, Dose 2 | 2.0 [1.0 to 4.0] | 7.0 [2.0 to 7.0]
  Myalgia, Overall: number analyzed (Participants) | 65 | 31
  Myalgia, Overall | 3.0 [1.0 to 4.0] | 5.0 [1.0 to 7.0]
  Shivering, Dose 1: number analyzed (Participants) | 10 | 13
  Shivering, Dose 1 | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 7.0]
  Shivering, Dose 2: number analyzed (Participants) | 23 | 9
  Shivering, Dose 2 | 1.0 [1.0 to 2.0] | 3.0 [2.0 to 7.0]
  Shivering, Overall: number analyzed (Participants) | 29 | 16
  Shivering, Overall | 1.0 [1.0 to 2.0] | 2.5 [1.0 to 7.0]
  Temperature, Dose 1: number analyzed (Participants) | 13 | 6
  Temperature, Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Temperature, Dose 2: number analyzed (Participants) | 21 | 7
  Temperature, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Temperature, Overall: number analyzed (Participants) | 31 | 13
  Temperature, Overall | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

6. Primary Outcome: Number of Subjects With Unsolicited Symptoms (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants
  At least one symptom | 51 | 44
  Subjects with grade 3 AEs | 7 | 5
  Subjects with related AEs | 7 | 3

7. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology
Time Frame: From first vaccination (Month 0) up to 1 month post last vaccination (Month 2).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants | 0 | 0

8. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongatoion of hospitalization, or result in disability /incapacity. Related = SAE assessed by the investigator as related to the vaccination.
Time Frame: From first vaccination (Month 0) up to 1 month post last vaccination (Month 2).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants
  Any SAEs | 6 | 5
  Related SAEs | 0 | 0

9. Primary Outcome: Number of Subjects With Renal Allograft Rejection
Description: Renal allograft rejection was confirmed through biopsy.
Time Frame: From the first vaccination (Month 0) up to 1 month post last vaccination (Month 2).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants
  Rejection confirmed | 0 | 0
  Rejection not confirmed | 0 | 3

10. Primary Outcome: Number of Subjects With Changes in Allograft Function
Description: Allograft function was indicated by the increase in levels of serum creatinine (≥ 1.20, ≥ 1.50, ≥ 1.75 or ≥ 2 fold increase). The number of subjects with declining allograft function, as determined by serum creatinine measurements post-vaccination (up to 30 days post-last vaccination) compared to pre-vaccination were presented.
Time Frame: From the first vaccination (Month 0) up to 1 month post last vaccination (Month 2).
Population: The analysis was performed on subjects with pre and post vaccination serum creatinine data available up to Month 2, from the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 113 | 107
Participants
  ≥1.20 fold increase | 5 | 7
  ≥1.50 fold increase | 0 | 1
  ≥1.75 fold increase | 0 | 1
  ≥2 fold increase | 0 | 1

11. Secondary Outcome: Anti-gE Antibody Concentrations
Description: Varicella Zoster Virus (VZV) gE antibody Immunoglobulin G concentrations were determined by ELISA assay, presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). The reference seropositivity cut-off value was ≥ 97 mIU/mL.
Time Frame: At Months 0, 1, 2, 7 and 13
Population: The analysis was performed on the adapted ATP cohort for humoral immunogenicity, which included all evaluable subjects up to Month 13, who did not meet any of the criteria for elimination from an ATP analysis, and for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 121 | 119
mIU/mL
  anti-gE, Month 0 | 1354.4 [1118.3 to 1640.4] | 1495.7 [1202.3 to 1860.8]
  anti-gE, Month 1 | 9530.5 [7111.3 to 12772.7] | 1501.9 [1231.3 to 1832.0]
  anti-gE, Month 2 | 19163.8 [15041.5 to 24416.0] | 1489.4 [1215.8 to 1824.7]
  anti-gE, Month 7: number analyzed (Participants) | 110 | 115
  anti-gE, Month 7 | 13066.7 [10291.5 to 16590.4] | 1533.7 [1249.6 to 1882.3]
  anti-gE, Month 13: number analyzed (Participants) | 111 | 111
  anti-gE, Month 13 | 8545.1 [6753.7 to 10811.5] | 1572.7 [1269.6 to 1948.1]

12. Secondary Outcome: Number of Subjects With a Vaccine Response for Anti-gE Humoral Immunogenicity
Description: Vaccine response was defined as: For initially seronegative subjects, antibody concentration at post-vaccination greater than or equal to (≥) 4 fold the cut-off for Anti-gE (4x97 mIU/mL); For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration. Vaccine response was determined by ELISA.
Time Frame: At Months 1, 7 and 13
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 121 | 119
Participants
  anti-gE, Month 1 | 77 | 3
  anti-gE, Month 7: number analyzed (Participants) | 110 | 114
  anti-gE, Month 7 | 83 | 5
  anti-gE, Month 13: number analyzed (Participants) | 111 | 109
  anti-gE, Month 13 | 74 | 7

13. Secondary Outcome: Frequencies of gE-specific Cluster of Differentiation 4 (CD4+) T-cells
Description: Descriptive statistics of gE-specific CD4+ T-cells, expressing at least two activation markers (from among interferon gamma [IFN-γ], interleukin-2 [IL-2], tumour necrosis factor alpha [TNF-α] and cluster of differentiation 40-ligand [CD40L]) were tabulated, as determined by in vitro Intracellular Cytokine Staining (ICS).
Time Frame: At Months 0, 2 and 13
Population: The analysis was performed on the adapted ATP cohort for cell-mediated immunogenicity (CMI), which included all evaluable subjects up to Month 13, who did not meet any of the criteria for elimination from an ATP analysis, and who were part of a CMI sub-cohort (Blood samples collected at Visits 1, 3 and 5 were analyzed to assess CMI response).
Measure: Mean (Standard Deviation); unit: gE-specific CD4+ T-cells/million T-cells
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 33 | 31
gE-specific CD4+ T-cells/million T-cells
  Month 0: number analyzed (Participants) | 31 | 30
  Month 0 | 110.9 (182.09) | 165.75 (242.92)
  Month 2: number analyzed (Participants) | 32 | 31
  Month 2 | 2433.07 (2102.29) | 156.98 (274.81)
  Month 13 | 1320.92 (1823.64) | 129.41 (197.92)

14. Secondary Outcome: Number of Subjects With a Vaccine Response for gE-specific CD4+ T-cells
Description: Vaccine response for gE-specific CD4+ T-cells expressing at least two activation markers (from among IFN-γ, IL-2, TNF-α and CD40L), was determined by in vitro ICS. Vaccine response was defined as: For initially subjects with pre-vaccination T-cell frequencies below the threshold, at least a 2-fold increase as compared to the threshold (2x<320> Events/10 million CD4+ T-cells); For initially subjects with pre-vaccination T-cell frequencies above the threshold, at least a 2-fold increase as compared to pre-vaccination T-cell frequencies.
Time Frame: At Months 2 and 13
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 30 | 28
Participants
  Month 2: number analyzed (Participants) | 28 | 28
  Month 2 | 20 | 0
  Month 13: number analyzed (Participants) | 30 | 27
  Month 13 | 17 | 0

15. Secondary Outcome: Number of Subjects With Any and Related SAEs
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related = SAE assessed by the investigator as related to the vaccination.
Time Frame: From 1 month post last vaccination (Month 2) until study end (Month 13).
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.If a subject reported a SAE exactly 1 month post-last vaccination (Month 2), it is possible that he/she might have also been taken into consideration for the Day0 up to Month2 SAEs assessment
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants
  Any SAEs | 21 | 29
  Related SAEs | 0 | 1

16. Secondary Outcome: Number of Subjects With Any pIMDs
Description: as for outcome 7
Time Frame: From 1 month post last vaccination (Month 2) until study end (Month 13).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants | 4 | 2

17. Secondary Outcome: Number of Subjects With Renal Allograft Rejection
Description: Renal allograft rejection was confirmed through biopsy.
Time Frame: From 1 month post last vaccination (Month 2) until study end (Month 13).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 132 | 132
Participants
  Rejection confirmed | 4 | 7
  Rejection not confirmed | 12 | 13

18. Secondary Outcome: Number of Subjects With Changes in Allograft Function
Description: Allograft function was indicated by the increase in levels of serum creatinine (≥ 1.20, ≥ 1.50, ≥ 1.75 or ≥ 2 fold increase). The number of subjects with declining allograft function, as determined by serum creatinine measurements post-vaccination (from 30 days post-last vaccination up to study end) compared to pre-vaccination were presented.
Time Frame: From 1 month post last vaccination (Month 2) until study end (Month 13)
Population: The analysis was performed on subjects with pre and post vaccination serum creatinine data available from Month 2 to Month 13, from the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 130 | 132
Participants
  ≥1.20 fold increase | 17 | 22
  ≥1.50 fold increase | 4 | 3
  ≥1.75 fold increase | 3 | 1
  ≥2 fold increase | 2 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period, Unsolicited symptoms: during the 30-day (Days 0-29) post-vaccination period, Serious Adverse Events: from Month 0 up to study end at Month 13.
Arm/Group | GSK1437173A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 1/132 | 1/132
Serious Adverse Events (participants affected / at risk) | 26/132 | 33/132
Other Adverse Events (participants affected / at risk) | 121/132 | 78/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=132) | Placebo Group (N=132)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 2 (2)
Transplant rejection (Immune system disorders) | 2 (2) | 4 (4)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 1 (1)
Renal graft infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (4)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=132) | Placebo Group (N=132)
Chills (General disorders) | 29 (33) | 16 (22)
Erythema (Skin and subcutaneous tissue disorders) | 33 (45) | 2 (2)
Fatigue (General disorders) | 62 (96) | 54 (79)
Gastrointestinal disorder (Gastrointestinal disorders) | 24 (31) | 24 (30)
Headache (Nervous system disorders) | 44 (68) | 35 (48)
Myalgia (Musculoskeletal and connective tissue disorders) | 65 (90) | 31 (42)
Pain (General disorders) | 114 (202) | 11 (14)
Pyrexia (General disorders) | 32 (37) | 14 (14)
Swelling (General disorders) | 15 (21) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.